CLINICAL TRIAL: NCT05102201
Title: National Tainan Junior College of Nursing
Brief Title: Effect of the Group-based Paro Intervention on Physiological and Psychological Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Tainan Junior College of Nursing (Other)
Responsible Party: Principal Investigator, Shu-Chuan Chen, 78, Sec. 2, Minzu Rd., West Central Dist., Tainan City 700007, Taiwan, R.O.C., National Tainan Junior College of Nursing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Shu-Chuan Chen
Record Dates: First submitted 2021-09-15; First posted 2021-11-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Dementia, Mild; Dementia Moderate; Cognitive Impairment
Keywords: Dementia; Paro; Neurobiology; Cognitive Function; Mental well-being
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Cognitive Dysfunction; Psychological Well-Being | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A randomized controlled trail, single-blind, two parallel groups, and repeated measures design
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation to treatment groups was concealed from participants until it was operationally required to begin intervention activities (ie, postbaseline data collection). Research assistants involved in data collection and data coding were masked to the other intervention groups through assignment of work to 1 group only, and by separate working locations. Intervention RAs were allocated to specific facilities, working with only one of the groups, and were masked to all outcome measurements, as were participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paro intervention group (Experimental): Participants in the Paro intervention group will receive a group (6-8 people as a group), facilitated, and 30-minute weekly session Paro intervention for 6 weeks.
  Interventions: Device: Paro (social robot) intervention
- control group (No Intervention): The control group will receive care as usual activities, such as painting, drawing, and craft, which are provided by each facility.

INTERVENTIONS:
Device: Paro (social robot) intervention — Participants in the Paro group will receive a group (6-8 people as a group), facilitated, and 30-minute weekly session Paro intervention for 6 weeks
  Arms: Paro intervention group

SUMMARY:
This project contains three studies. This study will use a pilot randomized controlled trial to examine the effect of Paro (social robot) intervention on oxytocin, dopamine, and HRV variations and mental well-being for specific attachment older adults with dementia. A randomized controlled trial, single-blind, two parallel groups, and repeated measures design were used to examine the effects of Paro intervention on neurobiologically changes and mental well-being for specific attachment older adults with dementia before, during, and after the intervention.

DETAILED DESCRIPTION:
This project contains three studies. Study 1 will use a randomized controlled trial to examine the effect of Paro (social robot) intervention on oxytocin, dopamine, and HRV variations for specific attachment older adults with dementia. A randomized controlled trial, single-blind, two parallel groups, and repeated measures design were used to examine the effects of Paro intervention on neurobiologically changes for specific attachment older adults with dementia before, during, and after the intervention. A sample of 120 older adults with dementia who are 65 years or older living in long-term care will be invited. Older adults will be randomly assigned to two groups: experimental group or control group. The outcomes will be assessed based on the change of dopamine and HRV at baseline, 3rd week during the Paro intervention, the end of intervention (6th week), and the 1 month after the Paro intervention. Furthermore, the change of oxytocin will be assessed at two time points: baseline and the end of Paro intervention. Study 2 will focus on the 60 participants of the 2 experimental groups. A mixed-method combined qualitative and quantitative research design will be used to explore the participating experience, group interaction, and its' association with mental health. Based on study 1 design, the outcomes of study 3 will be assessed based on the change of cognitive, executive functions, loneliness, depression, and well-being at the same points of study 1.

In addition, the Revised Adult Attachment Scale Chinese version (RAAS-C) will be used to classify the attachment types of the elderly. A sub-group analysis will be conducted to further understand the changes in the physical and mental health of the elderly with different attachment types after receiving Paro intervention. The results of this study will be used to provide empirical evidence to identify the effectiveness of Paro intervention on neurobiologically changes, cognition, executive functions, and mental well-being for older people with dementia. These results can be promoted as a care model in long-term facilities in the future.

ELIGIBILITY:
Inclusion Criteria:

(1) aged 65 years or over; (2) Mild to moderator dementia (3) an ability to communicate in Mandarin or Taiwanese; and (4) has been living in the LTC facility at least 3 months

Exclusion Criteria:

(1) have severe difficulty in communication; (2) are totally dependent on carers for daily activity; (3) have a diagnosed infectious disease, severe dementia, and severe mental illness such as schizophrenia and delusional disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Eligibility is based on gender which is a person's self-representation of gender identity.
Enrollment: 118 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Oxytocin | Change from Baseline Oxytocin at 6 weeks
  Blood samples for the oxytocin assay will collected from the antecubital vein into pre-chilled 5 ml EDTA tubes with 250 KIU of apoprotinin, and refrigerated until processing.
Finger tapping test (FTT) | Change from Baseline FTT at 6 weeks
  The FTT consists of tapping with the index finger on a computer mouse as many times as possible within 60 second.
HRV measurements | Change from Baseline HRV at 6 weeks
  It collects in this study using the Wireless Physiological Feedback System (Model NeXus 4) manufactured by Mind Media in the Netherlands. This device sets 400 signal acquisitions per minute and regularly corrects the device to maintain good reliability. Signal acquisition is managed, corrected, and heart rate frequency calculated by BioTrace+ software (Mind Media). Autonomic neuro physiological status reflect by the amplitude of high-frequency (HF) and low-frequency (LF) waveforms that were analyzed with the LF/HF ratio.
The Chinese version of Mini-Mental State Examination (MMSE) | Change from Baseline MMSE at 6 weeks
  The MMSE is a widely used tool that screens for levels of cognitive impairment, using the concepts of orientation, registration, attention and calculation, recall, and language. The MMSE score ranges from 0 to 30. In general, a cut-off point higher than 24 indicates normal cognition; 20-23 mild cognitive impairment; 10-19 moderate cognitive impairment; and 0-9 severe cognitive impairment.
Core components of executive functions- WM and response inhibition | Change from Baseline WM and response inhibition at 6 weeks
  The two core executive functions, WM and inhibition, were assessed using computerized tasks. Working memory was assessed using verbal WM and visuo-spatial WM tasks. Response inhibition was assessed using CWS, SS and GNG tasks.
Core components of executive functions- WM(1) -Verbal WM task | Change from Baseline Verbal WM task at 6 weeks
  Verbal WM task: These are powerpoint slides. Each slide has different numbers of red circles with squares as distracters. The task is to count the total number of red circles in each slide, keep the total in memory and recall the numbers in the correct order. The test starts with a length of memory recall (span) of two, that is, the participant had to recall two slides first. Each level of memory recall consists of three trials and the test is concluded when the participant failed two trials out of three at that same length of recall. If the participant is successful in 2 out of three trials, he/ she is allowed to go to the next span. A total score is calculated after adding a mark for each correct recall.
Core components of executive functions- WM(2)-Visuo-spatial WM task | Change from Baseline Verbal WM task at 6 weeks
  Visuo-spatial WM task: A 4 × 4 matrix with 16 squares is displayed on the computer screen as a pig house with a pig appearing in each window one at a time. The task is to recall in reverse order the locations where each target (pig) has appeared. The test start with a span length of two, that is, two pigs appear one after another. Each span consist of two trials and the test is concluded when the participant failed both trials at that same span length. Each correct location is given one point with a maximum score of 88. The score is taken as the measure of Visuo-spatial WM. At the end of the test, obtain score is automatically displayed on the computer screen.
Core components of executive functions- response inhibition (1)-Color word Stroop task | Change from Baseline Color word Stroop task at 6 weeks
  Color word Stroop task: In this task different colour words will appear on the computer screen one at a time. The task is to name the color the word is printed, disregarding what the color word reads. The colour of the word printed is in the same color as the meaning of the word (congruent trials, eg; "red" is printed in red colour), or it is different from the meaning (incongruent trials, eg; word "green" is printed in blue colour). There are 75 congruent trials and 25 incongruent trials for one test session. Incorrect responses on incongruent trials are taken to assess the level of inhibitory control. The higher the errors the lower the interference control is.
Core components of executive functions- response inhibition (2)-Stop signal task | Change from Baseline Stop signal task at 6 weeks
  Stop signal task: It assess the ability to inhibit ongoing responses. This is like a car game where a car appears on the computer screen. Every time the car appear, the participant is supposed to press a designated key as fast as possible to drive the car away. But when a stop-sign board appeared next to the car, participants has to refrain from pressing for the car to stand still. Each session in this task consist of 24 trials with six stop-signs-trials. Number of incorrect presses in stop sign (commission errors) is considered as the measure of inhibition and it is automatically displayed on the screen at the end of the task.
Core components of executive functions- response inhibition (3)-Go/no-go task | Change from Baseline Go/no-go task at 6 weeks
  Go/no-go task (two versions: colour and shape): It assess ability to inhibit pre potent responses. The subject is presented with four different stimuli on the screen, one at a time in random order. There are two squares and two circles in blue and red. In the first session, the subject is instructed to respond by pressing a key each time when a blue figure appeared (go-trials) regardless of the shape, and not to respond when a red figure appear. In the second session, the subject is instructed to respond each time when a square appear, regardless of the color, and not to respond when a circle appear. Together the two consecutive sessions include 60 stimuli with 77% go-trials. The number of incorrect responses (commission errors) is used as a measure of inhibition and it is automatically displayed on the screen at the end of the task.
Geriatric Depression Scale - Short Form (GDS-SF) | Change from Baseline GDS-SF at 6 weeks
  The GDS-SF consists of 15 items with 10 positive items and 5 negative items and has been found to be a useful tool to detect depressive symptoms in older populations. The scores range from 0-21 and a cut-off point of 6 or more indicates the presence of depression.
The UCLA Loneliness Scale version 3 (UCLA-3) | Change from Baseline UCLA-3 at 6 weeks
  The UCLA loneliness is used to measure a person's subjective feelings of loneliness and feelings of isolation. Each item on the scale is rated from 1 (Never) to 4 (Often) with a total score ranging from 20 to 80. The scale does not identify a cut-off score that defines loneliness. The higher the score, the more severe a person's feelings of loneliness.
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Change from Baseline WEMWBS at 6 weeks
  The WEMWBS scale was developed by researchers at the Universities of Warwick and Edinburgh (2006), including 14 items of mental well-being covering subjective well-being and psychological functioning. The scale is scored by summing responses to each item answered on a 5 points Likert scale and the scores range from 14 - 70. The higher the score, the better the mental well-being.

SECONDARY OUTCOMES:
Group atmosphere | week-1, week-3 and week-10
  The Chinese version of the group climate questionnaire, 12 items, was developed by Zhong et al. (2013). This questionnaire consists three main dimensions including engagement (5 items), conflict (3 items), and avoidance (4 items). Each item on the scale is rated from 1 (Never) to 4 (Often) with a total score ranging from 12 to 48. The scale does not identify a cut-off score that defines good or bad group climate. The higher the score, the more better group atmosphere participant perceived.
Group satisfaction | week-1, week-3 and week-6
  The group satisfaction scale was developed Keyton (1991). The Chinese version of group satisfaction scale, which consists 14 items, was translated and modified by Lin. This questionnaire consists five main dimensions including group process feelings, attitudes of leaders, attitudes of group members, group acceptance, group equality. Each item on the scale is rated from 1 (very satisfied) to 5 (very dissatisfied) with a total score ranging from 14 to 70.The higher the score, the more dissatisfied the group is.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital Dou-Liou Branch, Douliu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
IPD Sharing Access Criteria may be shared

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT05102201/Prot_SAP_000.pdf